CLINICAL TRIAL: NCT05319847
Title: An Exploratory Investigation of a Male Focused Skincare Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Let's Disco (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20239Disco
Record Dates: First submitted 2022-03-31; First posted 2022-04-08 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Acne; Skin Abnormalities
MeSH Terms: conditions — Acne Vulgaris; Skin Abnormalities

STUDY DESIGN:
Masking Description: Open Label, Single Group Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Daily Skin Supplement - Fountain of Youth
  Interventions: Dietary Supplement: Daily Skin Supplement - Fountain of Youth

INTERVENTIONS:
Dietary Supplement: Daily Skin Supplement - Fountain of Youth — Skincare supplement

SUMMARY:
Most skincare products on the market are topical and do not take a holistic approach to understanding skin health. This trial will examine a dietary supplement designed to support the gut microbiome and promote skin health from an internal perspective. Research has previously supported the link between the gut microbiome and skin health and the supplement tested in this trial will further the knowledge on the effectiveness of supporting gut health to improve skin outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Between the ages of 18-55
* Frequently experience different forms of acne
* Frequently experience breakouts
* Must be in good health with no long term health conditions
* BMI must be under 40
* Must follow a consistent dietary regimen
* Must be willing to stop any oral supplementation targeting their skin while in the trail

Exclusion Criteria:

* Anyone who does take prescription medication (oral or topical) targeting their skin including reinoid, over the counter retinol, or retinal
* Not willing to stop any oral supplementation targeting their skin
* Severe chronic conditions, including oncological and psychiatric disorders
* Previous severe allergic reactions
* Unwilling the follow the study protocol

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 38 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Adult Acne | 12 week
  Change in overall frequency and intensity of adult acne (Likert Scale 0-5 with higher scores representing a reduction in the appearance of adult acne)

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided